CLINICAL TRIAL: NCT05821998
Title: Effect of Thoracic Block Technique on Arterial Blood Gases, Vital Signs and Lung Compliance in Children With Atelectasis on Mechanical Ventilation
Brief Title: Effect of Thoracic Block Technique on Arterial Blood Gases in Children With Atelectasis on Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Abdallah Amin, Scientific researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P. T. REC/012/004401
Record Dates: First submitted 2023-03-25; First posted 2023-04-20 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Atelectasis; Intensive Care Unit; Children
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic block technique and designed chest physical therapy program (Experimental): Manual compression on healthy lung for 20 seconds and rest for 20 seconds, total time 20 minutes and percussion, vibration and modified postural drainage on session time for 35 minutes every day for ten days
  Interventions: Other: Thoracic block technique
- Designed chest physical therapy program (Active Comparator): Percussion, vibration and modified postural drainage for 30 minutes every day for ten days
  Interventions: Other: Designed chest physical therapy program

INTERVENTIONS:
Other: Thoracic block technique — Manual compression of the healthy lung during expiration associated with the use of invasive or non invasive mechanical ventilation
  Other Names: Technique of insufflation to reverse atelectasis
  Arms: Thoracic block technique and designed chest physical therapy program
Other: Designed chest physical therapy program — Percussion, vibration and modified postural drainage
  Arms: Designed chest physical therapy program

SUMMARY:
Statement of the problem:

• Does the thoracic block technique has effect on arterial blood gases, vital signs and lung compliance in children with atelectasis on mechanical ventilation? Null hyposis there is no effect of thoracic block technique on arterial blood gases, vital signs and lung compliance in children with atelectasis on mechanical ventilation.

DETAILED DESCRIPTION:
Subjects:

The study targets the children from both sexes.diagnosed with atelectasis in intensive care unit. Sample size estimation will be carried out to determine the recruited number of children, selected randomly from Cairo University pediatric specialized hospital, Cairo to participate in the study,

Study design:

Randomized controlled clinical trial. Children will receive intervention type randomly, 22 child received percussion, vibration, modified postural drainage and the other 22 child will receive percussion, vibration, modified postural drainage and thoracic block technique.

Children will be assessed by measuring heart rate, respiratory rate,which reflect the physiological status, arterial blood gases which include partial pressure of oxygen (PaO2), partial pressure of carbon dioxide (PaCO2) and oxygen saturation (SaO2) and dynamic lung compliance which reflect clinical improvement of chest condition before and after ten days of receiving intervention

ELIGIBILITY:
Inclusion Criteria:

1. age range from 4 months to 4 years.
2. diagnosed with pneumonia, receiving mechanical ventilation.
3. start from second day of admission to intensive care unit
4. have unilateral mild to moderate atelectasis according to medical referral.
5. should be vitally stable during the session.

Exclusion Criteria:

The children were excluded from the study if they had one of the following:

1. medically unstable ( examples: tachycardia and tachypnea)
2. uncontrolled convulsion.
3. rib fracture.
4. pneumothorax -

Ages: 4 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment of oxygenation status | 10 days for each participant
  Assessment of change of partial pressure of arterial oxygen which is one value in arterial blood gases test results which calculated by arterial blood gases analyzier and comparing results before and after intervention
Assessment of ventilation status | 10 days for each participant
  Assessment of change of partial pressure of carbon dioxide which is one value of arterial blood gases test results and calculated by arterial blood gases analyzier before and after intervention
Assessment of dynamic lung compliance | 10 days for each participant
  Assessment of change in lung compliance value during air flow which calculated automatically by mechanical ventilator, we record it before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Abdallah, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt